CLINICAL TRIAL: NCT03062839
Title: Melatonin as Adjuvant Treatment for ADHD in Adults
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hospital Israelita Albert Einstein (Other)
Collaborators: Fundação de Amparo à Pesquisa do Estado de São Paulo (Other Government); University of Sao Paulo (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: TDAHMEL
Record Dates: First submitted 2017-02-20; First posted 2017-02-23 (Actual); Last update posted 2018-08-15 (Actual); Status verified 2018-07

CONDITIONS: Attention Deficit Hyperactivity Disorder
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity | interventions — Melatonin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Melatonin (Experimental): Melatonin 5 mg taken 30 minutes before bed time
  Interventions: Drug: Melatonin 5 mg
- Placebo (Placebo Comparator): Placebo identical to melatonin capsule taken 30 min before bed time
  Interventions: Drug: Melatonin 5 mg

INTERVENTIONS:
Drug: Melatonin 5 mg — Melatonin 5 mg taken 30 minutes before bed time
  Other Names: Melatonina

SUMMARY:
This study aims to evaluate the effect of melatonin supplementation as adjuvant treatment in ADHD in adults.

ELIGIBILITY:
Inclusion Criteria:

Male and female age 18-60 inclusive. Primary diagnosis of ADHD AISRS total score ≥ 24 CGI-S ≥4 (moderately ill or worse). Understands and is able, willing, and likely to fully comply with the study procedures and restrictions.

Has given written informed consent to participate in the study.

Exclusion Criteria:

BMI less than18.5 or greater than 35. Any underlying/ history or current diagnosis of systemic and/or metabolic disease (e.g. diabetes, Crohn's disease) and/or neurological condition state that may render the subject illegible to participate in the study as assessed by medical history, physical exam, clinical and lab evaluation.

History of uncontrolled hypertension or a resting systolic blood pressure > 140mmHg or diastolic blood pressure > 90mmHg (Subjects with well controlled hypertension on a stable dose (2 months) of anti-hypertensives will be allowed to participate).

Major depression or anxiety disorder which is a focus of treatment or requires taking medication.

A lifetime history of psychosis or bipolar disorder Has any concurrent chronic or unstable medical condition that could confound with the results of safety assessments, increase risk to the subject or lead to difficulty complying with the protocol.

Subjects taking any medication with CNS effects Subjects with a history of two or more prior failed adequate trials of ADHD treatment due to adverse events.

Use of dietary supplements with potential CNS effect, including omega-3 supplements, 30 days before study initiation and throughout the study.

Clinical history of cognitive impairment in judgment of investigator. Pregnant or breast-feeding subjects. Women of childbearing potential must have a negative pregnancy test performed at screening visit prior to randomization. Women of childbearing potential must agree to use adequate birth control for the entire duration of the study.

Subjects with a current (within the last 3 months) DSM-V diagnosis of alcohol or drug abuse or dependence (excluding nicotine).

Has taken an investigational drug or taken part in a clinical trial within 30 days prior to screening.

Any other reason that, in the opinion of the investigator, prevents the subject from participating in the study or compromise the subject safety.

Previous use of melatonin or melatonin analogues

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 120 (Estimated)
Dates: Start 2017-09-01 (Actual); Primary Completion 2019-02-28 (Estimated); Study Completion 2019-06-30 (Estimated)

PRIMARY OUTCOMES:
Adult ADHD Investigator Symptom Rating Scale. | 12 weeks
  Each of the individual DSM-IV symptoms of ADHD is rated 0 to 3 on a scale of severity.

SECONDARY OUTCOMES:
Anxiety | 12 weeks
  GAD-7 scale
Depression | 12 weeks
  PHQ-9 scale
CGI-S / I | 12 weeks
  Clinical Global Impression Severity / Improvement
Adverse Event Monitoring | 12 weeks
  Adverse Event Monitoring

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital Albert Einstein, São Paulo, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: No